CLINICAL TRIAL: NCT00150605
Title: A Phase IIIb, Open Label Observational Study of SPD417 Used in Combination With Other Psychotropic Medications for the Treatment of Bipolar I Disorder
Brief Title: Safety of SPD417 Combined With Other Psychotropic Medications in the Treatment of Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Validus Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD417-308
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2007-11-02 (Estimated); Status verified 2006-06

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

INTERVENTIONS:
Drug: Extended-release carbamazepine

SUMMARY:
The purpose of this study is to evaluate the safety of SPD417 when given with other psychotropic medications to treat bipolar I disorder.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria for Bipolar I disorder
* Screening YMRS score =>16
* Women of childbearing potential agree to take adequate precautions against contraception
* Currently receiving treatment with antipsychotic therapy or combination therapy of mood stabilizer and antipsychotic

Exclusion Criteria:

* Hospitalization required for treatment of psychiatric symptoms
* Patients who meet DSM-IV for ultra-rapid cycling
* History of serious suicide attempt requiring medical intervention
* Female subjects who are pregnant or lactating, including females with a positive pregnancy test at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-02; Study Completion 2005-10

PRIMARY OUTCOMES:
Safety as assessed by treatment-emergent adverse events over 8 weeks of treatment

SECONDARY OUTCOMES:
YMRS Scale
Clinical Global Impressions Scale - Bipolar Version
HAM-D and MADRS Scales for Depression